CLINICAL TRIAL: NCT00780169
Title: A Phase I Study of Sorafenib (Nexavar®) in Combination With FOLFIRI as First Line Therapy for Metastatic Colorectal Cancer
Brief Title: Phase I Trial of Sorafenib + FOLFIRI In Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTT 06-08
Record Dates: First submitted 2008-10-23; First posted 2008-10-27 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sorafenib +FOLFIRI (Experimental): This is a Phase I safety study. There is only one arm of FOLFIRI administered every 14 days (2 week schedule) and sorafenib administered orally, twice daily continuously. First cycle sorafenib began at day +2 to FOLFIRI.
  Interventions: Drug: sorafenib + FOLFIRI

INTERVENTIONS:
Drug: sorafenib + FOLFIRI — escalating doses of sorafenib and irinotecan
  * sorafenib starting dose 400 mg/day
  * irinotecan starting dose 80 mg/m2 on day 1
  Other Names: sorafenib - Nexavar

SUMMARY:
The purpose of this study is to assess the safety, the maximum tolerated dose and the recommended dose for phase II studies of a chemotherapy-combination of sorafenib, irinotecan, and 5-fluorouracil (5-FU)/folinic acid (FA) (FOLFIRI) as first-line treatment for metastatic colorectal cancer.

DETAILED DESCRIPTION:
A standard phase I dose escalation design with three to six patients per dose level will be used. The first three patients will receive chemotherapy at the dose level 1 for 4 weeks (2 FOLFIRI regimen). The dose will be escalated for the next patients by one dose level if none of the three patients at a dose level experience a dose-limiting toxicity (DLT) during the first six weeks. Intrapatient dose escalation is not allowed. If one of the three patients has a DLT, an additional three patients will be enrolled at this dose level and the dose will be escalated if no additional patients experience a DLT. Otherwise, the dose escalation will be stopped, and the last dose will be regarded as the Maximum Administered Dose (MAD). The preceding dose level will be declared the Maximum Tolerated Dose (MTD). This dose level will be the recommended dose (RD). At least 6 patients will be treated at the MTD. The cohort at the MTD dose level can be expanded to as many as 12 patients to gain experience with the toxicities and efficacy of Sorafenib + FOLFIRI combination over a broad patient range. Patients experiencing a DLT during the first cycle of treatment will have the drug withheld. They will be eligible for repeated treatment at a lower dose or treated off protocol.

Treatment is to be discontinued in cases of serious or unmanageable toxicity or request by the patient. Otherwise therapy will continue until clinically or radiologically documented disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal cancer
* Histopathological verification of the primary tumor
* Measurable disease according to RESIST criteria
* Response Evaluation Criteria in Solid Tumors (ECOG) performance status ≤ 2
* Age > 18 years.
* Women of childbearing potential must have had a negative pregnancy test within 7 days prior to start of treatment. Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.
* Patients may have had prior adjuvant chemotherapy with fluoropyrimidines WITHOUT pelvic radiotherapy.
* Radiation: Patients may have had prior palliative radiation therapy to NO more than 50% of the areas bearing of bone marrow stores.
* Adequate organ and marrow function : Hemoglobin > 9.0 g/dl; absolute neutrophil count (ANC) >1,500/mm3; absolute granulocyte count(AGC) > 1.5 x 109 /L; Platelets > 100 x 109 /L; Serum creatinine and creatinine clearance within upper normal limit; Bilirubin < 1.0 x upper normal limit, < 2.5 x upper normal limit if documented liver metastases; aspartate aminotransferase (AST) < 2.5 x upper normal limit, < 5 x upper normal limit if documented liver metastases
* Life expectancy > 3 months
* Informed consent

Exclusion Criteria:

* Previous or concurrent malignancies
* Patients with central nervous system (CNS) metastases
* Pregnant or lactating women
* Concurrent treatment with other experimental drugs or anticancer therapy
* Previous chemotherapy for advanced and/or metastatic disease
* Previous adjuvant therapy with irinotecan or targeted agents
* Previous Sorafenib therapy
* Previous full dose curative pelvic radiotherapy
* History of cardiovascular disease, cerebral ischemia infarction or hemorrhage, Gilbert's disease, HIV positivity
* Unable to be compliant with the procedures in the protocol
* Currently use prohibited medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-10; Primary Completion 2011-05 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Toxicity spectrum of Sorafenib (MTD, DLT) and the recommended dose (RD) for phase II studies of Sorafenib when combined with FOLFIRI in first line patients with metastatic colorectal cancer (mCRC) | each cycle - 4 weeks; continuous monitoring of AEs

SECONDARY OUTCOMES:
Pharmacokinetics of Irinotecan in the presence of Sorafenib | 2 years
Response according to Response Evaluation Criteria in Solid Tumors (RECIST) | every 2 cycles - 8 weeks
Time to Progression and Overall Survival | each cycle - 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean A Maroun, MD, Principal Investigator — The Ottawa Hospital Regional Cancer Centre
Locations (1):
- The Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada